CLINICAL TRIAL: NCT00721461
Title: Probe Study of the Tolerability of an Investigational Electroporation Device, MedPulser (Trademark) DNA Delivery System (DDS) in Healthy Adults 18 to 35 Years of Age
Brief Title: A Study to Test the Tolerability of an Investigational Electroporation Device in Healthy Adults (V930-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: University of California, San Diego (Other); Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: V930-001; 2008_537
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: Assess; Tolerability; MedPulser DDS device

ARMS (1):
- 1 (Experimental): V930
  Interventions: Biological: V930

INTERVENTIONS:
Biological: V930 — Intramuscular injection of phosphate buffered saline solution will be given and within 2 - 5 minutes will be followed by an electrostimulation pulse with the MedPulser DDS in the deltoid muscle of the right arm. 15 days later, the same procedure will take place using the left arm.

SUMMARY:
A study to evaluate the tolerability of electrostimulation applications with an investigational device known as the MedPulser DDS.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18 and 35
* Woman who are able to become pregnant must use an acceptable form of birth control

Exclusion Criteria:

* You are breast feeding
* You have taken any type of pain reliever within 12 hours of electrostimulation
* You have participated in another clinical study within 4 weeks of starting this study or plan to participate in another clinical study while participating in this study
* You have muscle atrophy, weakness or neuromuscular disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Assess the tolerability of the MedPulser DDS device. | Severity of pain will be measured at time of treatment and 1, 5, 10, and 20 minutes and 24 hours after electrostimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC